CLINICAL TRIAL: NCT04109651
Title: Influence of Nursing Intervention on Mother and Infant, Materna Attachment, Parental Self-efficacy, Infant Development
Brief Title: The Effect of Nursing Interventions on Maternal Attachment, Parental Self-efficacy and Infant Development
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KTO Karatay University (Other)
Responsible Party: Principal Investigator, Figen Türkdüdükçü, Teaching a-Assistant, KTO Karatay University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: KaratayU
Record Dates: First submitted 2019-09-25; First posted 2019-09-30 (Actual); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Nurse's Role; Parenting; Self Efficacy; Development, Child; Attachment
MeSH Terms: interventions — Methods

STUDY DESIGN:
Intervention Model Description: Interventional (Clinical Trial)
Who Masked: Outcomes Assessor
Masking Description: The last data were collected nurses from primary health center (not researher) who did not know anything about participants of experiment and control group.
  Data recorded on the computer by the assistant investigator without specifying the experiment and control group.
  The experimental and control groups codified by the co-investigator. The analysis of the data encoded by the groups was done by a statistical expert. Data collectors, statistical analyzes and report writing were blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nursing İntervention (Experimental): Intervention: Other: Nursing intervention
  Interventions: Other: Nursing intervention
- No Intervention: Control Group (Other): Receive routine nursing care
  Interventions: Other: Nursing intervention

INTERVENTIONS:
Other: Nursing intervention — Nursing Intervention: This intervention was planned based on Meleis' Transition Theory. So it includes individual counseling and training.
  In the Health Promotion Monitoring Program; three training modules and one reminder module were implemented and telephone counseling was provided. Various training tools were used in these trainings. Three different power point presentations were made during the training sessions. Illustrated printed training material was used. At the end of the training, training booklet was given to the participants.
  Other Names: No Intervention: Control Group

SUMMARY:
The aim of this study was to determine the effects of Meleis 'Transition Theory based health improvement monitoring program on infants' development, maternal attachment and parental self-efficacy in 36-40 weeks of gestation and in the first and fourth months after birth. Sample was 64 (experimental group:32; control group: 32), alfa=0,05 and power=0.80 at the end of study. The experimental group received nursing interventions based on Meleis' Transition Theory, while the control group received routine primary health care. Data were collected 3 times: pretest, 3 and 7 months after intervention (for experimental group) and 3 and 7 months after pretest (for control group).

DETAILED DESCRIPTION:
Motherhood is one of the most important milestones in a woman's life, and at the same time the beginning of a process in which very important responsibilities are undertaken. The mother needs knowledge, skills and energy to fulfill her new responsibilities. The development of motherhood identity is the process of learning motherhood behaviors of women. This process starts with the recognition of pregnancy, develops during pregnancy and continues after birth. Transition Theory is a suitable tool for nurses to understand the transition to parenting, a developmental type of transition. Appropriate nursing interventions tailored to the needs of pregnant women and women who have just given birth are needed. Targeted / predicted change in the large / large effect size of the mothers in the experimental group (effect size 0.80, 80% of the standard deviation) with the Health Promotion Monitoring Program, the sample calculation with 5% alpha error and 80% power was the minimum for each group. It was determined that a total of 52 people (26 *) should be recruited (G * Power 3.1.9.2). It was decided to include at least 32 people in each working group with a 20% surplus, considering that they might be lost in data collection. Women's experiences in transition to motherhood should be sought to propose, define, and explain professional interventions. In this study, a Health Promotion Program starting from 36-40 weeks of gestation until the sixth month of birth was administered to the mothers registered at the primary health care center in Karatay, Konya. In this study, the investigator planned to increase maternal infant attachment, to increase parental self-efficacy, to keep infant development at the best level, thus ensuring a healthy transition for the mother.

Duration of intervention and collecting data for the study was 11 months. Data was collected using information form (21 item; information about participant, parents and infant), three scales (Turkish Version of Maternal Attachment Inventory; parental self-efficacy scale, Denver II development screening test). Scales validation and reliability studies were made for Turkish population.

ELIGIBILITY:
Inclusion Criteria:

* Having at least primary school graduation
* 18 Years and older
* Lack of any chronic disease

Exclusion Criteria:

* Multiple pregnancy
* Risk of preterm birth
* Does not speak Turkish
* Pregnant / mothers not attending at least one education and / or measurement
* Want to leave the work
* Presence of mental or physical illnesses such as postpartum depression during follow-up
* Baby; Presence of congenital and / or metabolic disease during prenatal and postnatal postnatal follow-up

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 64 (Actual)
Dates: Start 2018-10-03 (Actual); Primary Completion 2019-08-12 (Actual); Study Completion 2019-08-12 (Actual)

PRIMARY OUTCOMES:
infant development level | At the end of 7 month
  infant development at a high level

SECONDARY OUTCOMES:
Maternal attachment scores | At the end of 7 month
  Mother will increase infant attachment level
Parental self-efficacy scales scores | At the end of 7 month
  Mother self-efficacy level will increase

CONTACTS AND LOCATIONS:
Overall Officials: FATMA TAŞ ARSLAN, Study Director — SELÇUK UNİVERSİTY
Locations (1):
- Kto Karatay University, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I do not plan to share any data of participants.